CLINICAL TRIAL: NCT04305210
Title: Alzheimer's Disease: Clinical Investigation and Neuroimage Studies Including 18F-PM-PBB3 and 18F-florbetapir (AV-45) PET Examination
Acronym: PMPBB3/AV45
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201802170A0
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; mild cognitive impairment; Neuroimages; 18F-PM-PBB3; 18F-flobetapir (AV-45); PET; MRI; Tau protein; Amyloid
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Frontotemporal Dementia | interventions — florbetapir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-18-PMPBB3 (Experimental): F-18-PMPBB3 imaging
  Interventions: Drug: F-18 PMPBB3
- 18F-florbetapir (Experimental): 18F-florbetapir (AV45) imaging
  Interventions: Drug: 18F-florbetapir

INTERVENTIONS:
Drug: F-18 PMPBB3 — In this study we will enroll 20 healthy controls, 20 amnestic mild cognitive impairment patients (aMCI), 20 mild-moderate dementia due to AD patients and 10 other dementia such as frontotemporal dementia patients. All of the subjects will receive 18F-PM-PBB3 tau PET scan, and 18F-flobetapir (AV-45) amyloid PET scan, brain magnetic resonance images and clinical evaluation.
  Arms: F-18-PMPBB3
Drug: 18F-florbetapir — 18F-florbetapir
  Arms: 18F-florbetapir

SUMMARY:
Dementia is a common neurodegenerative syndrome in aged population. Alzheimer's disease (AD) is the most common disease. The main pathological findings in AD include senile plaques (SP) and neurofibrillary tangles (NFT). The b-amyloid is the main peptide in SP and tau protein is the main finding in NFT. In addition, b-amyloid is considered as a disease biomarker, but the severity of AD is related with the tau protein.

Recently a new tracer 18F-PM-PBB3 has been introduced in tau PET images. In a prelimary study with the 18F-PM-PBB3, the tau PET scan provide a good tool to evaluate tau deposition pattern among healthy volunteers, and patients with mild and moderate dementia due to AD. In this study we will enroll 20 healthy controls, 20 amnestic mild cognitive impairment patients (aMCI), 20 mild-moderate dementia due to AD patients and 10 other dementia such as frontotemporal dementia patients. All of the subjects will receive 18F-PM-PBB3 tau PET scan, and 18F-flobetapir (AV-45) amyloid PET scan, brain magnetic resonance images and clinical evaluation. We will follow up the clinical features for 2 years to understand the disease progression, disease conversion from aMCI to AD.

The study aims to investigate the deposition patterns of tau protein with 18F-PM-PBB3 and amyloid protein with 18F-flobetapir in patients with amnestic mild cognitive impairment due to AD, mild to moderate degree of dementia due to AD and healthy controls. The study will provide the information of these two proteins in different stages of dementia patients. The results may help the strategy in selection of anti-dementia drugs in the pharmaceutical company and industry and reduce the economic burden for the society. The study also can improve the understanding of Alzheimer's disease in academic research.

ELIGIBILITY:
Inclusion Criteria:

* Patient with probable AD (Appendix I) Inclusion criteria

  1. Age ranges from 45~90 years
  2. Patients fulfill the criteria of probable AD (DSM IV and NINCDS-ADRDA)
  3. Mild cognitive impairment to moderate dementia (CDR: 0.5 to 2.0 or MMSE: 10-25)
  4. Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study

Patient with amnestic MCI due to AD criteria (Appendix II: criteria proposed by world ADNI) Inclusion criteria

1. Age ranges from 45~90 years
2. Patients fulfill the criteria of aMCI (The early aMCI and late aMCI were proposed by world ADNI)
3. Amnestic mild cognitive impairment (CDR: 0.5 or MMSE: 26-30, with logical memory >=7)
4. Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study

Patients with probable FTD (Appendix III) 1, 2, 3 Inclusion criteria

1. Age ranges from 45~90 years
2. Patients fulfill the criteria of probable FTD
3. Mild cognitive impairment to moderate dementia (CDR: 0.5 to 2.0 or MMSE: 10-25)
4. Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study

Healthy control Inclusion criteria

1. Age ranges from 45~90 years
2. Normal cognitive function (CDR: 0 or MMSE: 26-30)
3. Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study

Exclusion Criteria:

* 1) Implantation of metal devices including cardiac pacemaker, intravascular metal devices.

  2) Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases 3) Major psychiatric disorders, drug or alcohol abuse and major depression 4) Pregnant women or breast- feeding women 5) Subjects in whom MRI was contraindicated 6) History of severe allergic or anaphylactic reactions particularly to the tested drugs 7) History of positive test for human immunodeficiency virus (HIV) 8) Indication of impaired liver function as shown by an abnormal liver function profile at screening (eg. repeated values of aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≧ 3X the upper limit of normal values)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-01-23 (Estimated); Study Completion 2021-01-23 (Estimated)

PRIMARY OUTCOMES:
Tau Distribution | 1 YEAR
  Tau Distribution Among healthy controls, amnestic mild cognitive impairment patients (aMCI), mild-moderate dementia due to AD and other dementia such as frontotemporal dementia. Subjects Measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-PM-PBB3 tau PET Scan and AV45 amyloid pet scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan District, Guishan Dist,, Taiwan